CLINICAL TRIAL: NCT05888480
Title: Effects of a Culturally Specific End-of-life Communication Skills Training for Chinese Oncology Nurses
Brief Title: A Culturally Specific End-of-life Communication Skills Training
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: The Hong Kong Polytechnic University (Other)
Responsible Party: Principal Investigator, Dr Joyce Chung, Assistant Professor, School of Nursing, The Hong Kong Polytechnic University
Allocation: Randomized | Model: Sequential | Masking: Double | Purpose: Other
Other Study IDs: HSEARS20230525002
Record Dates: First submitted 2023-02-09; First posted 2023-06-05 (Actual); Last update posted 2024-02-28 (Actual); Status verified 2024-02

CONDITIONS: End-Of-Life
Keywords: Communication; Nurse; Terminally ill
MeSH Terms: conditions — Death; Communication

STUDY DESIGN:
Intervention Model Description: The IG will receive the end-of-life CST between the two measurement points, and the CG will be a waitlist group and receive the training after the end of data collection.
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention group (IG) (Experimental): The IG will receive the end-of-life CST between the two measurement points
  Interventions: Other: The end-of-life communication skills training
- Control group (CG) (Other): The CG will be a waitlist group and receive the training after the end of data collection.
  Interventions: Other: Routine training activity

INTERVENTIONS:
Other: The end-of-life communication skills training — Training methods include lectures, video demonstrations, and simulation in small groups (4-5 trainees per group with multidisciplinary roles). Written and audiovisual learning materials will be offered. Each session will be 150 minutes, including lectures and video demonstration (90 min/session) and simulation and feedback (60 min/session). One session will be conducted in two weeks. Totally there will be four sessions completed in 8 weeks.
  Arms: Intervention group (IG)
Other: Routine training activity — Routine training activities arranged by relevant departments in hospitals
  Arms: Control group (CG)

SUMMARY:
The goal of this clinical trial is to evaluate the effectiveness of culturally specific end-of-life communication skills training (CST) among Chinese oncology nurses.

The main question it aims to answer is: What is the effectiveness of culturally specific end-of-life CST among Chinese oncology nurses? Participants will receive an 8-week communication skills training. Researchers will compare the intervention group and the wait-list group to see if skills, self-efficacy, and outcome expectancy beliefs will be improved.

DETAILED DESCRIPTION:
Objectives: The study aims to evaluate the effectiveness of culturally specific end-of-life CST among Chinese oncology nurses.

Design and participants: It is designed as a single-blind, pre-post randomized controlled trial (RCT). Registered nurses who work with advanced cancer patients in hospital settings will be recruited. The participants will be randomly assigned to either the intervention group (IG) or the control group (CG). The IG will receive the end-of-life CST between the two measurement points, and the CG will be a waitlist group and receive the training after the end of data collection.

Data analysis: Demographic information about the participants will be summarised in descriptive statistics. Independent t-tests and chi-square tests are used to investigate the comparability of groups in terms of the demographics generated by randomization. The primary and secondary outcome variables will be examined using covariate-adjusted linear mixed models. This approach enables the consideration of missing data. For non-repeated continuous measurements, ordinary linear regression and logistic models will be adopted. The intention-to-treat (ITT) analysis and post hoc analyses of contaminated data will be performed.

Expected results: Nurses' skills, self-efficacy, and outcome expectancy beliefs will improve after the CST.

ELIGIBILITY:
Inclusion Criteria:

* Registered nurses who work with advanced cancer patients in hospital settings
* Consent to participate in the study

Exclusion Criteria:

* Nurses working temporarily in the two hospitals as scholars or trainees from other hospitals
* Specialized nurses in palliative care

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 148 (Estimated)
Dates: Start 2023-09-01 (Actual); Primary Completion 2024-10 (Estimated); Study Completion 2024-12 (Estimated)

PRIMARY OUTCOMES:
Change from Baseline Skills at 3 months | up to 3 months
  Measured by Nurses' Clinic Communication Competency Scale, a 58-item self-reported scale which measures six dimensions. A 5-point Likert scale from (1) very poor to (5) very good is used. Higher scores mean a better outcome.

SECONDARY OUTCOMES:
Change from Baseline Self-efficacy at 3 months | up to 3 months
  Measured by Hospice Care Self-efficacy Scale on nurses, a 12 items with a 5-point Likert scale from (1) very diffident to (5) very confident. Higher scores mean a better outcome.
Change from Baseline Outcome expectancy beliefs 3 months | up to 3 months
  Measured by The Communication Outcomes Questionnaire, a 23-item self-report questionnaire with a 9-point Likert scale from 1 = very likely and 9 = very unlikely. Higher scores mean a worse outcome.

OTHER OUTCOMES:
Acceptance and satisfaction | up to 3 months
  Self-developed items and open questions anout the training experience

CONTACTS AND LOCATIONS:
Overall Officials: Joyce Chung, PhD, Principal Investigator — The Hong Kong Polytechnic University
Locations (1):
- Zhejiang Cancer Hospital, Hangzhou, Zhejiang, China

IPD SHARING:
Plan to Share IPD: No